CLINICAL TRIAL: NCT06029296
Title: Proof of Concept: Diclofenac as a KMO Inhibitor in Individuals With Alcohol Use Disorder
Brief Title: Diclofenac as a KMO Inhibitor
Acronym: DKMOI
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Daniel Roche, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HP-00107035
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder
Keywords: diclofenac
MeSH Terms: conditions — Alcoholism | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diclofenac (Active Comparator): Participants will take a single 100mg dose of diclofenac.
  Interventions: Drug: Diclofenac
- Placebo (Placebo Comparator): Participants will take a single dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac — 100 mg
  Arms: Diclofenac
Drug: Placebo — Sugar pill
  Arms: Placebo

SUMMARY:
This mechanistic, proof of concept laboratory study will test the pharmacological properties of diclofenac in individuals with AUD. Participants will complete two sessions in which they will receive a single dose of diclofenac (100 mg) or matched placebo in a randomized and double blind fashion. The primary aim is to assess whether this dose of diclofenac, vs. placebo, increases circulating levels of kynurenic acid. This finding would provide evidence that diclofenac (100 mg) inhibits the kynurenine 3-monooxygenase enzyme.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-65
* Meet DSM-5 diagnostic criteria for AUD of any severity (Mild, Moderate, or Severe)

Exclusion Criteria:

* Lifetime DSM-5 diagnosis of schizophrenia spectrum and other psychotic disorders and bipolar and related disorders
* Positive urine toxicology screen for the following substances: cocaine, opiates, amphetamines, methamphetamine, phencyclidine, barbiturates, benzodiazepine, methadone, and tricyclic antidepressants
* Self-reported daily use of opioids (including prescribed)
* Serious alcohol withdrawal symptoms as indicated by a score ≥ 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised
* If female: pregnant, nursing, or with reproductive potential who refuses to use reliable methods of birth control throughout the study
* Any autoimmune disorder, inflammatory disorder, or medical condition that may interfere with safe study participation and/or study aims (e.g., any cardiac, renal, or liver disease, uncontrolled hypertension, or diabetes)
* Attempted suicide in the past 3 years and/or serious suicidal intention or plan within the past year
* Currently on prescription medication that contraindicates use of diclofenac, including but not necessarily limited to: oral corticosteroids, anticoagulants, lithium, warfarin, aspirin (daily use), methotrexate, cyclosporine, ACE-inhibitors, and diuretics like furosemide and thiazides
* Previously known hypersensitivity, including gastroenteritis, asthma, and allergic-type reactions, to any NSAID and/or aspirin
* Current daily use of any NSAID or regular pattern of near daily use within the past three months, regular use of a prebiotic or probiotic supplement and/or any antibiotic, prebiotic, or probiotic use within the last month
* Any lifetime history of ulcer disease, gastritis, gastroenteritis, or gastrointestinal bleeding
* Current or recent (within 3 months) participation in a clinical trial involving medication administration
* Currently in treatment, a history of treatment within the 30 days before enrollment, or currently seeking immediate treatment for AUD
* Current (last 12 months) DSM-5 diagnosis of SUD for any psychoactive substances other than alcohol and nicotine
* Currently prescribed a psychotropic medication for the treatment of schizophrenia spectrum and other psychotic disorders, bipolar and related disorders
* AST and ALT > four times the upper limit of the normal range, or albumin, GFR, BUN, or creatinine 15% > the upper limit of the normal range
* Suffered a mild or moderate traumatic brain injury (TBI) within the last 12 months, a severe TBI at any point in their life, or a moderate TBI before the age of 12
* Has below a 6th grade reading level
* Within the last 3 months, tested positive for COVID-19 (i.e. the SARS-CoV-2 virus) and experienced common related symptoms
* Any other circumstances that, in the opinion of the investigators, compromises participant safety, ability of the investigators to conduct the study as designed, and/or study integrity

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Kynurenic Acid | 0-, 60-, 120-, 180-, and 240-minutes after pill administration
  Serum levels of Kynurenic Acid

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roche, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Maryland Psychiatric Research Center (MPRC) Treatment Research Program (TRP), Catonsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No